CLINICAL TRIAL: NCT00968071
Title: A Phase II Study of Decitabine and Gemtuzumab Ozogamicin in Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Decitabine and Gemtuzumab Ozogamicin in Acute Myelogenous Leukemia and High-risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0882
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Leukemia; AML; MDS; High-Risk Myelodysplastic Syndrome; Decitabine; 5-aza-2 deoxycytidine; Dacogen; Gemtuzumab Ozogamicin; Mylotarg
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Decitabine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine + Gemtuzumab Ozogamicin (Experimental): Decitabine 20 mg/m^2 intravenously (IV) over an hour and half daily for 5 days, Gemtuzumab Ozogamicin 3 mg/m^2 IV on day 5.
  Interventions: Drug: Decitabine; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Decitabine — 20 mg/m^2 IV over an hour and half daily for 5 days.
  Other Names: Dacogen
Drug: Gemtuzumab Ozogamicin — 3 mg/m^2 IV on day 5.
  Other Names: Gemtuzumab; Mylotarg

SUMMARY:
The goal of this clinical research study is to learn if giving 5-aza-2 deoxycytidine (decitabine) in combination with Mylotarg (gemtuzumab ozogamicin) can help to control AML or high-risk MDS. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Gemtuzumab ozogamicin is designed to attach to Sialic acid-binding Ig-like lectin 3 (CD33), a certain protein that is often found in leukemia cells, causing them to die.

Decitabine is designed to damage the DNA (the genetic material) of cells, which may cause cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive decitabine through a needle in your vein over 1 and 1/2 hours on Days 1-5 of each cycle. You will also receive gemtuzumab ozogamicin by vein over about 1 hour after you receive decitabine on Day 5 of each 4-6 week cycle.

During Cycle 1 only, if a bone marrow test done 2 weeks after you receive your first study drug treatment shows abnormal leukemia cells, you will receive another treatment with decitabine intravenously over 1 and 1/2 hours for 5 days.

Gemtuzumab may cause allergic reactions, nausea, and vomiting. To help prevent such side effects, you will receive Benadryl (diphenhydramine) and hydrocortisone. You may receive these drugs by vein, or by mouth on the days you get gemtuzumab ozogamicin during the entire study.

Study Visits:

During Cycle 1, blood (about 2 teaspoons) will be drawn at least 1 time each week for routine tests. If the doctor thinks it is necessary, you may be asked to have additional blood drawn.

During Cycle 1, after approximately 2 weeks of your first study drug administration , you will have a bone marrow aspiration to decide whether you will receive additional decitabine in Cycle 1.

During Cycles 2-3, blood (about 2 teaspoons) will be drawn for routine tests at least 2 times each month.

During Cycles 4 and beyond, blood (about 2 teaspoons) will be drawn for routine tests at least 1 time each month.

If the doctor thinks it is necessary, you may have a bone marrow aspirate every 1 to 3 months to check the status of the disease.

Length of Study:

You may receive the combination of decitabine and gemtuzumab ozogamicin for up to 6 cycles. After this, if your doctor thinks it is in your best interest, you may continue to take decitabine alone for up to 24 cycles. You will be taken off study early if the disease gets worse, you experience intolerable side effects, or your doctor thinks that it is no longer in your best interest to receive the study drug(s).

Long-term Follow-up:

Once you are off study, you will have follow up visits every month for up to 2 years. At these visits, blood (about 2 teaspoons) will be drawn for routine tests.

This is an investigational study. Gemtuzumab ozogamicin is FDA approved and commercially available for the treatment of AML that has come back after treatment in patients over the age of 65 years. Decitabine is FDA approved and commercially available for the treatment of MDS. The use of gemtuzumab ozogamicin and decitabine in combination is investigational.

Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >/= to 16 years at the time of signing the informed consent form.
3. Diagnosis of Acute myeloid leukemia (AML) [other than acute promyelocytic leukemia (APL)] with refractory/relapsed disease. Patients with newly diagnosed AML will be eligible if not a candidate for intensive chemotherapy. Patients with high-risk Intermediate-2 or high by International Prognostic Scoring System (IPSS) or >/= to 10% blasts) MDS will also be eligible. All non-hematological toxicity of previous cancer therapy should have resolved to </= grade 1 (except alopecia or other toxicities not involving major organs).
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= to 3 at study entry.
5. Laboratory test results within these ranges (unless due to leukemia): Serum creatinine </= 2 mg/dL Total bilirubin </= 2 mg/dL aspartate aminotransferase (AST) (SGOT) and/or alanine aminotransferase (ALT) (SGPT) </= 2.5 x ULN or </= 5 times Upper limit of normal (ULN) if related to disease
6. Women of childbearing potential (WCBP) must have a negative urine pregnancy test within 7 days and must either commit to continued abstinence from heterosexual intercourse or adopting at least one highly effective method of contraception. These methods include intra-uterine device, tubal ligation, partner's vasectomy, hormonal birth control pills. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk.
3. Use of any other experimental drug or therapy for leukemia within 7 days unless there is clear evidence of rapid disease progression.
4. Use of hydrea to control proliferative disease will be allowed prior to starting therapy on study and for up to 7 days each during cycle 1-3 (Maximum daily dose of 7gm).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2/19/2008 through 5/12/2009. All participants recruited at UT MD Anderson Cancer Center.
Groups:
- Decitabine + Gemtuzumab Ozogamicin: Decitabine 20 mg/m^2 intravenously (IV) over an hour and half daily for 5 days plus Gemtuzumab Ozogamicin 3 mg/m^2 IV on day 5.
Period: Overall Study
Arm/Group | Decitabine + Gemtuzumab Ozogamicin
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Decitabine Gemtuzumab Ozogamicin: Decitabine 20 mg/m^2 IV over an hour and half daily for 5 days Plus Gemtuzumab Ozogamicin 3 mg/m^2 IV on day 5.
Arm/Group | Decitabine Gemtuzumab Ozogamicin
Number analyzed (Participants) | 71
Age Continuous [Median (Full Range); unit: years] | 65 [26 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: Complete Response (CR) was defined as normalization of peripheral blood and bone marrow with </= 5% blasts, a peripheral anc >/= 1 * 10^9 /l, and a platelet count of >/= 100 & 10^9 /l. Evaluation after each treatment course (5-6 weeks) up to 6 cycles.
Time Frame: Up to 36 weeks
Measure: Number; unit: participants
Arm/Group | Decitabine Gemtuzumab Ozogamicin
Number analyzed (Participants) | 71
participants | 3

ADVERSE EVENTS:
Time Frame: Four years, six months
Arm/Group | Decitabine Gemtuzumab Ozogamicin
Serious Adverse Events (participants affected / at risk) | 15/71
Other Adverse Events (participants affected / at risk) | 44/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine Gemtuzumab Ozogamicin (N=71)
Death (General disorders) | 15 (15)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine Gemtuzumab Ozogamicin (N=71)
Infection other (Infections and infestations) | 22 (24)
Febrile Neutropenia (Infections and infestations) | 24 (27)
Hemorrhage (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes